CLINICAL TRIAL: NCT01631552
Title: A Phase I/II Study of IMMU-132 (hRS7-SN38 Antibody Drug Conjugate) in Patients With Epithelial Cancer
Brief Title: Study of Sacituzumab Govitecan-hziy (IMMU-132) in Adults With Epithelial Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMMU-132-01
Record Dates: First submitted 2012-06-26; First posted 2012-06-29 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Gastric Adenocarcinoma; Esophageal Cancer; Hepatocellular Carcinoma; Non-small Cell Lung Cancer; Small Cell Lung Cancer; Ovarian Epithelial Cancer; Carcinoma Breast Stage IV; Hormone-refractory Prostate Cancer; Head and Neck Cancers- Squamous Cell; Renal Cell Cancer; Urinary Bladder Neoplasms; Cervical Cancer; Endometrial Cancer; Glioblastoma Multiforme; Triple Negative Breast Cancer; Pancreatic Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Ovarian Epithelial; Breast Neoplasms; Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Glioblastoma; Triple Negative Breast Neoplasms; Pancreatic Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sacituzumab Govitecan-hziy (SG) 8 mg/kg (Experimental): Participants will receive sacituzumab govitecan-hziy (SG) 8 mg/kg of body weight via intravenous (IV) infusion on Days 1 and 8 of a 21-day treatment cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Sacituzumab Govitecan-hziy (SG)
- SG 10 mg/kg (Experimental): Participants will receive SG 10 mg/kg of body weight via intravenous (IV) infusion on Days 1 and 8 of a 21-day treatment cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Sacituzumab Govitecan-hziy (SG)
- SG 12 mg/kg (Experimental): Participants will receive SG 12 mg/kg of body weight via intravenous (IV) infusion on Days 1 and 8 of a 21-day treatment cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Sacituzumab Govitecan-hziy (SG)
- SG 18 mg/kg (Experimental): Participants will receive SG 18 mg/kg of body weight via intravenous (IV) infusion on Days 1 and 8 of a 21-day treatment cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Sacituzumab Govitecan-hziy (SG)

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy (SG) — Administered via intravenous (IV) infusion
  Other Names: hRS7-SN38; IMMU-132

SUMMARY:
The primary objective in Phase I is to evaluate the safety and tolerability of sacituzumab govitecan-hziy (SG) as a single agent administered in 21-day treatment cycles in previously treated participants with advanced epithelial cancer. In Phase II, the primary objective is to evaluate the safety and efficacy of sacituzumab govitecan-hziy administered in 21-day treatment cycles at a dose selected in Phase I.

Tumor types in the study will include: cervical, colorectal, endometrial, ovarian, esophageal, gastric adenocarcinoma, glioblastoma multiforme, head and neck cancers- squamous cell, hepatocellular, prostate, non-small-cell lung cancer, pancreatic, renal cell, small-cell lung cancer, non-triple negative breast cancer (non-TNBC), triple-negative breast cancer (TNBC) and metastatic urothelial cancer (mUC).

DETAILED DESCRIPTION:
The outcome measures are planned to be assessed up to the data cutoff date. Following the data cutoff date, the participants will either stay on the study and will be followed for safety data collection or rolled into another Gilead-sponsored study. Therefore, only safety data will be collected after the data cutoff date.

ELIGIBILITY:
Inclusion Criteria:

* Individuals able to understand and give written informed consent.
* Histologically or cytologically confirmed epithelial cancer of one of the following types:

  * Gastric adenocarcinoma (GC)
  * Esophageal cancer (EC)
  * Hepatocellular carcinoma (HCC)
  * Non-small-cell lung cancer (NSCLC)
  * Small-cell lung cancer (SCLC)
  * Epithelial ovarian cancer (EOC)
  * Cervical Cancer
  * Endometrial Cancer
  * Triple-negative breast cancer (TNBC)
  * Non-triple-negative breast cancer
  * Papillary thyroid cancer (excludes follicular, medullary, Hurthle cell, and anaplastic thyroid cancer)
  * Glioblastoma multiforme (GBM)
  * Hormone-refractory prostate cancer (HRPC)
  * Head and neck cancers- squamous cell (SCCHN)
  * Renal cell cancer (clear cell) (RCC)
  * Urothelial cancer
  * Stage IV (metastatic) disease (except for individuals with GBM).
* Refractory to or relapsed after at least one prior standard therapeutic regimen
* Adequate performance status (ECOG 0 or 1)
* Expected survival ≥ 6 months.
* Measurable disease by CT or MRI.
* At least 2 weeks beyond treatment (chemotherapy, investigational drugs including small molecular inhibitors, immunotherapy and/or radiation therapy) or major surgery and recovered from all acute toxicities to Grade 1 or less (except alopecia).
* At least 2 weeks beyond high dose systemic corticosteroids (however, low dose corticosteroids < 20 mg prednisone or equivalent daily are permitted).
* Adequate hematology without ongoing transfusional support (hemoglobin > 9 g/dL, absolute neutrophil count (ANC) > 1,500 per mm^3, platelets > 100,000 per mm^3).
* Adequate renal and hepatic function (creatinine ≤ 2.0 x institutional upper limit of normal (IULN), bilirubin ≤ 1.5 IULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x IULN or 5 x IULN if know liver metastases).
* Otherwise, all toxicity at study entry ≤ Grade 1.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Women of childbearing potential and fertile men unwilling to use effective contraception during study until conclusion of 12-week post-treatment evaluation period.
* Individuals with Gilbert's disease.
* Individuals with brain metastases can be enrolled only if treated, non-progressive brain metastases and off high-dose steroids (> 20 mg prednisone or equivalent) for at least 4 weeks.
* Presence of bulky disease (defined as any single mass > 7 cm in its greatest dimension). Individuals with a mass over 7 cm, but otherwise eligible, may be considered for enrollment after discussion and approval with the medical monitor.
* Individuals with active ≥ grade 2 anorexia, nausea or vomiting, and/or signs of intestinal obstruction.
* Individuals with non-melanoma skin cancer or carcinoma in situ of the cervix are eligible, while individuals with other prior malignancies must have had at least a 3-year disease-free interval.
* Individuals known to be HIV positive, hepatitis B positive, or hepatitis C positive.
* Known history of unstable angina, MI, or CHF present within 6 months or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring anti-arrhythmia therapy.
* Known history of clinically significant active COPD, or other moderate-to-severe chronic respiratory illness present within 6 months.
* Prior history of clinically significant bleeding, intestinal obstruction, or GI perforation within 6 months of initiation of study treatment.
* Infection requiring intravenous antibiotic use within 1 week.
* History of an anaphylactic reaction to irinotecan or ≥ Grade 3 GI toxicity to prior irinotecan,
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2012-12-17 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (12):
- United States (12):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Helen F. Graham Cancer Center, Newark, Delaware
  - MD Anderson Cancer Center Orlando (UF Health Cancer Center), Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - IU Health Goshen Cancer Center, Goshen, Indiana
  - Massachusettes General Hospital, Boston, Massachusetts
  - Weill Cornell/New York Presbyterian Hospital, New York, New York
  - Columbia University Herbert Irving Cancer Center, New York, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology Sammons Cancer Center, Dallas, Texas
  - Virginia Mason Cancer Center, Seattle, Washington

REFERENCES:
- [Result] Kalinsky K, Diamond JR, Vahdat LT, Tolaney SM, Juric D, O'Shaughnessy J, Moroose RL, Mayer IA, Abramson VG, Goldenberg DM, Sharkey RM, Maliakal P, Hong Q, Goswami T, Wegener WA, Bardia A. Sacituzumab govitecan in previously treated hormone receptor-positive/HER2-negative metastatic breast cancer: final results from a phase I/II, single-arm, basket trial. Ann Oncol. 2020 Dec;31(12):1709-1718. doi: 10.1016/j.annonc.2020.09.004. Epub 2020 Sep 15. PMID 32946924
- [Result] Santin AD, Komiya T, Goldenberg DM, et al. Sacituzumab govitecan (SG) in patients (pts) with previously treated metastatic endometrial cancer (mEC): results from a phase 1/2 study. J Clin Oncol. 2020; 38 (suppl; abstr 6081)
- [Result] Bardia A, Mayer IA, Kalinsky K. Sacituzumab Govitecan-hziy in Triple-Negative Breast Cancer. Reply. N Engl J Med. 2019 Jun 13;380(24):2382. doi: 10.1056/NEJMc1903943. No abstract available. PMID 31189049
- [Result] Bardia A, Mayer IA, Vahdat LT, Tolaney SM, Isakoff SJ, Diamond JR, O'Shaughnessy J, Moroose RL, Santin AD, Abramson VG, Shah NC, Rugo HS, Goldenberg DM, Sweidan AM, Iannone R, Washkowitz S, Sharkey RM, Wegener WA, Kalinsky K. Sacituzumab Govitecan-hziy in Refractory Metastatic Triple-Negative Breast Cancer. N Engl J Med. 2019 Feb 21;380(8):741-751. doi: 10.1056/NEJMoa1814213. PMID 30786188
- [Result] Tagawa ST, Faltas M, Lam ET, et al. Sacituzumab govitecan (IMMU-132) in patients with previously treated metastatic urothelial cancer (mUC): Results from a phase I/II study. J Clin Oncol. 2019;39(suppl 7S):abstr 354.
- [Result] Bardia A, Diamond JR, Vahdat LT, et al. Efficacy of sacituzumab govitecan (anti-Trop-2-SN-38 antibody-drug conjugate) for treatment-refractory hormone-receptor positive (HR+)/HER2- metastatic breast cancer (mBC). J Clin Oncol. 2018;36(15 suppl):1004.
- [Result] Gray JE, Heist RS, Starodub AN, Camidge DR, Kio EA, Masters GA, Purcell WT, Guarino MJ, Misleh J, Schneider CJ, Schneider BJ, Ocean A, Johnson T, Gandhi L, Kalinsky K, Scheff R, Messersmith WA, Govindan SV, Maliakal PP, Mudenda B, Wegener WA, Sharkey RM, Goldenberg DM. Therapy of Small Cell Lung Cancer (SCLC) with a Topoisomerase-I-inhibiting Antibody-Drug Conjugate (ADC) Targeting Trop-2, Sacituzumab Govitecan. Clin Cancer Res. 2017 Oct 1;23(19):5711-5719. doi: 10.1158/1078-0432.CCR-17-0933. Epub 2017 Jul 5. PMID 28679770
- [Result] Ocean AJ, Starodub AN, Bardia A, Vahdat LT, Isakoff SJ, Guarino M, Messersmith WA, Picozzi VJ, Mayer IA, Wegener WA, Maliakal P, Govindan SV, Sharkey RM, Goldenberg DM. Sacituzumab govitecan (IMMU-132), an anti-Trop-2-SN-38 antibody-drug conjugate for the treatment of diverse epithelial cancers: Safety and pharmacokinetics. Cancer. 2017 Oct 1;123(19):3843-3854. doi: 10.1002/cncr.30789. Epub 2017 May 30. PMID 28558150
- [Result] Heist RS, Guarino MJ, Masters G, Purcell WT, Starodub AN, Horn L, Scheff RJ, Bardia A, Messersmith WA, Berlin J, Ocean AJ, Govindan SV, Maliakal P, Mudenda B, Wegener WA, Sharkey RM, Goldenberg DM, Camidge DR. Therapy of Advanced Non-Small-Cell Lung Cancer With an SN-38-Anti-Trop-2 Drug Conjugate, Sacituzumab Govitecan. J Clin Oncol. 2017 Aug 20;35(24):2790-2797. doi: 10.1200/JCO.2016.72.1894. Epub 2017 May 26. PMID 28548889
- [Result] Bardia A, Mayer IA, Diamond JR, Moroose RL, Isakoff SJ, Starodub AN, Shah NC, O'Shaughnessy J, Kalinsky K, Guarino M, Abramson V, Juric D, Tolaney SM, Berlin J, Messersmith WA, Ocean AJ, Wegener WA, Maliakal P, Sharkey RM, Govindan SV, Goldenberg DM, Vahdat LT. Efficacy and Safety of Anti-Trop-2 Antibody Drug Conjugate Sacituzumab Govitecan (IMMU-132) in Heavily Pretreated Patients With Metastatic Triple-Negative Breast Cancer. J Clin Oncol. 2017 Jul 1;35(19):2141-2148. doi: 10.1200/JCO.2016.70.8297. Epub 2017 Mar 14. PMID 28291390
- [Result] Sharkey RM, McBride WJ, Cardillo TM, Govindan SV, Wang Y, Rossi EA, Chang CH, Goldenberg DM. Enhanced Delivery of SN-38 to Human Tumor Xenografts with an Anti-Trop-2-SN-38 Antibody Conjugate (Sacituzumab Govitecan). Clin Cancer Res. 2015 Nov 15;21(22):5131-8. doi: 10.1158/1078-0432.CCR-15-0670. Epub 2015 Jun 23. PMID 26106073
- [Result] Starodub AN, Ocean AJ, Shah MA, Guarino MJ, Picozzi VJ Jr, Vahdat LT, Thomas SS, Govindan SV, Maliakal PP, Wegener WA, Hamburger SA, Sharkey RM, Goldenberg DM. First-in-Human Trial of a Novel Anti-Trop-2 Antibody-SN-38 Conjugate, Sacituzumab Govitecan, for the Treatment of Diverse Metastatic Solid Tumors. Clin Cancer Res. 2015 Sep 1;21(17):3870-8. doi: 10.1158/1078-0432.CCR-14-3321. Epub 2015 May 5. PMID 25944802
- [Derived] Kwapisz D. Sacituzumab Govitecan-hziy in Breast Cancer. Am J Clin Oncol. 2022 Jul 1;45(7):279-285. doi: 10.1097/COC.0000000000000919. Epub 2022 May 12. PMID 35728046
- [Derived] Bardia A, Messersmith WA, Kio EA, Berlin JD, Vahdat L, Masters GA, Moroose R, Santin AD, Kalinsky K, Picozzi V, O'Shaughnessy J, Gray JE, Komiya T, Lang JM, Chang JC, Starodub A, Goldenberg DM, Sharkey RM, Maliakal P, Hong Q, Wegener WA, Goswami T, Ocean AJ. Sacituzumab govitecan, a Trop-2-directed antibody-drug conjugate, for patients with epithelial cancer: final safety and efficacy results from the phase I/II IMMU-132-01 basket trial. Ann Oncol. 2021 Jun;32(6):746-756. doi: 10.1016/j.annonc.2021.03.005. Epub 2021 Mar 16. PMID 33741442
- [Derived] Faltas B, Goldenberg DM, Ocean AJ, Govindan SV, Wilhelm F, Sharkey RM, Hajdenberg J, Hodes G, Nanus DM, Tagawa ST. Sacituzumab Govitecan, a Novel Antibody--Drug Conjugate, in Patients With Metastatic Platinum-Resistant Urothelial Carcinoma. Clin Genitourin Cancer. 2016 Feb;14(1):e75-9. doi: 10.1016/j.clgc.2015.10.002. Epub 2015 Oct 19. PMID 26541586
- [Derived] Cardillo TM, Govindan SV, Sharkey RM, Trisal P, Arrojo R, Liu D, Rossi EA, Chang CH, Goldenberg DM. Sacituzumab Govitecan (IMMU-132), an Anti-Trop-2/SN-38 Antibody-Drug Conjugate: Characterization and Efficacy in Pancreatic, Gastric, and Other Cancers. Bioconjug Chem. 2015 May 20;26(5):919-31. doi: 10.1021/acs.bioconjchem.5b00223. Epub 2015 May 8. PMID 25915780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 17 December 2012. The last study visit occurred on 13 August 2020.
  Outcome Measures were assessed up to the data cutoff date of 01 March 2019. Following the data cutoff date, the participants either stayed on the study and were followed for safety data collection or rolled into another Gilead-sponsored study. Therefore, only safety data was collected after the data cutoff date.
Pre-assignment Details: Tumor types included in the study were as follows: cervical, colorectal, endometrial, ovarian, esophageal, gastric adenocarcinoma, glioblastoma multiforme, head and neck cancers- squamous cell, hepatocellular, prostate, non-small-cell lung cancer, pancreatic, renal cell, small-cell lung cancer, non-triple negative breast cancer (non-TNBC), triple-negative breast cancer (TNBC) and metastatic urothelial cancer (mUC).
Groups:
- Sacituzumab Govitecan-hziy (SG) 8 mg/kg: Participants received sacituzumab govitecan-hziy (SG) 8 mg/kg of body weight via intravenous (IV) infusion on Days 1 and 8 of a 21-day treatment cycle until disease progression or unacceptable toxicity.
- SG 10 mg/kg: Participants received sacituzumab govitecan-hziy 10 mg/kg of body weight via IV infusion on Days 1 and 8 of a 21-day treatment cycle until disease progression or unacceptable toxicity.
- SG 12 mg/kg: Participants received sacituzumab govitecan-hziy 12 mg/kg of body weight via IV infusion on Days 1 and 8 of a 21-day treatment cycle until disease progression or unacceptable toxicity.
- SG 18 mg/kg: Participants received sacituzumab govitecan-hziy 18 mg/kg of body weight via IV infusion on Days 1 and 8 of a 21-day treatment cycle until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Sacituzumab Govitecan-hziy (SG) 8 mg/kg | SG 10 mg/kg | SG 12 mg/kg | SG 18 mg/kg
Started | 83 | 420 | 9 | 3
Enrolled and Treated | 81 | 402 | 9 | 3
Completed | 81 | 400 | 9 | 3
Not Completed | 2 | 20 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SG 8mg/kg: Participants received sacituzumab govitecan-hziy 8 mg/kg of body weight via IV infusion on Days 1 and 8 of a 21-day treatment cycle until disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | SG 8mg/kg | SG 10 mg/kg | SG 12 mg/kg | SG 18 mg/kg | Total
Number analyzed (Participants) | 81 | 402 | 9 | 3 | 495
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (10.91) | 59.8 (11.28) | 59.1 (10.53) | 56.0 (4.00) | 60.0 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 281 | 6 | 1 | 334
  Male | 35 | 121 | 3 | 2 | 161
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 67 | 329 | 6 | 3 | 405
  Race: Black | 6 | 19 | 2 | 0 | 27
  Race: Asian | 4 | 13 | 1 | 0 | 18
  Race: Other | 4 | 41 | 0 | 0 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 4 | 16 | 0 | 0 | 20
  Ethnicity: Not Hispanic or Latino | 77 | 386 | 9 | 3 | 475

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Any Treatment Emergent Adverse Events and Serious Treatment Emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) were defined as any adverse events (AEs) that begin or worsen on or after the start of study drug through 30 days after the last dose of study drug. The severity was graded based on the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 4.03. An AE that met one or more of the following outcomes was classified as serious:
  * Fatal
  * Life-threatening
  * Disabling/incapacitating
  * Results in hospitalization or prolongs a hospital stay
  * A congenital abnormality
  * Other important medical events may also be considered serious AEs if they may require medical or surgical intervention to prevent one of the outcomes listed above
  Per planned analysis, populations to be used for evaluation of this outcome measure were as follows: Triple Negative Breast Cancer (TNBC) Target Population, HR+/HER2- Metastatic Breast Cancer (mBC) Population, Metastatic Urothelial Cancer (mUC) Population, and Overall Safety Population.
Time Frame: First dose date up to last dose for data cutoff date of 01 March 2019 (maximum duration: 55.2 months) plus 30 days
Population: * Target mTNBC: Participants with mTNBC who received at least 2 prior therapies for metastatic disease & who received at least 1 dose of 10 mg/kg SG
  * HR+/HER2-mBC: Participants with HR+/HER2- mBC who progressed on at least 1 prior hormonal therapy & who received at least 1 dose of 10 mg/kg SG
  * mUC: Participants who had relapsed after or were refractory to at least 1 prior treatments & who received at least 1 dose of 10 mg/kg SG
  * OSP: All participants who received at least 1 dose of SG
Measure: Number; unit: Percentage of participants
Groups:
- TNBC Target Population: Overall 144 participants with TNBC were enrolled in the study and received at least one dose of SG. Of these 144 participants, 108 received at least 2 prior therapies for metastatic disease and were treated with SG at a starting dose of 10mg/kg. These 108 participants were included in the analysis of safety and were referred to as the TNBC Target Population.
- HR+/HER2- mBC Population: Overall 68 participants with non-TNBC were enrolled in the study and received at least one dose of SG. Of these 68 participants, 54 were confirmed as Hormone receptor-positive/Human epidermal growth factor receptor 2-negative (HR+/HER2-), had progressed on at least one prior hormonal therapy in the metastatic setting, and had received at least one dose of 10 mg/kg SG. These 54 participants were included in the analysis of safety and were referred to as the HR+/HER2- mBC Population.
- mUC Population: Overall 49 participants with metastatic urothelial cancer were enrolled in the study and received at least one dose of SG. Of these 49 participants, 45 had either relapsed after or were refractory to at least one prior standard therapeutic regimen and received at least one dose of 10 mg/kg SG. These 45 participants were included in the analysis of safety and were referred to as the mUC Population.
- Overall Safety Population (OSP): Overall 495 participants were enrolled in the study and received at least one dose of 10 mg/kg, 8 mg/kg, 12mg/kg, or 18mg/kg SG. These participants were included in the Overall Safety Population and analyzed for safety.
Arm/Group | TNBC Target Population | HR+/HER2- mBC Population | mUC Population | Overall Safety Population (OSP)
Number analyzed (Participants) | 108 | 54 | 45 | 495
Percentage of participants
  Adverse Events | 100.0 | 100.0 | 100.0 | 99.8
  Serious Adverse Events | 30.6 | 35.2 | 42.2 | 38.8

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Sacituzumab Govitecan-hziy (SG) Due to Any Adverse Events, Excluding Adverse Events Leading to Death
Description: Per planned analysis, populations to be used for evaluation of this outcome measure were as follows: Triple Negative Breast Cancer (TNBC) Target Population, HR+/HER2- Metastatic Breast Cancer (mBC) Population, Metastatic Urothelial Cancer (mUC) Population, and Overall Safety Population (OSP).
Time Frame: First dose date up to last dose for data cutoff date of 01 March 2019 (maximum duration: 55.2 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- HR+/HER2- mBC Population: Overall 68 participants with non-TNBC were enrolled in the study and received at least one dose of SG. Of these 68 participants, 54 were confirmed as HR+/HER2-, had progressed on at least one prior hormonal therapy in the metastatic setting, and had received at least one dose of 10 mg/kg SG. These 54 participants were included in the analysis of safety and were referred to as the HR+/HER2- mBC Population.
Arm/Group | TNBC Target Population | HR+/HER2- mBC Population | mUC Population | Overall Safety Population (OSP)
Number analyzed (Participants) | 108 | 54 | 45 | 495
Percentage of participants | 2.8 | 5.6 | 15.6 | 8.1

3. Primary Outcome: Percentage of Participants Who Required Dose Interruption Due to Any Adverse Events
Description: as for outcome 2
Time Frame: First dose date up to last dose for data cutoff date of 01 March 2019 (maximum duration: 55.2 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TNBC Target Population | HR+/HER2- mBC Population | mUC Population | Overall Safety Population (OSP)
Number analyzed (Participants) | 108 | 54 | 45 | 495
Percentage of participants | 45.4 | 46.3 | 51.1 | 51.7

4. Primary Outcome: Objective Response Rate (ORR) by Independent Central Review (ICR)
Description: ORR was defined as the rate an overall best response of either complete response (CR) or partial response (PR) by ICR assessment according to RECIST1.1. CR was defined as the disappearance of all target lesions and reduction in short axis of any pathologic lymphnode to <10 mm. PR was defined as ≥ 30% decrease in the sum of diameters of target lesions, taking the baseline sum diameters. Per planned analysis, ORR by ICR was assessed for the TNBC Target Population only.
Time Frame: Up to data cutoff date of 01 March 2019 (maximum duration: 74 months)
Population: Target mTNBC: Participants with mTNBC who received at least 2 prior therapies for metastatic disease and who received SG at a dose of 10 mg/kg.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TNBC Target Population
Number analyzed (Participants) | 108
Percentage of participants | 34.3 [25.4 to 44.0]

5. Primary Outcome: Objective Response Rate by Local Assessment
Description: ORR was defined as the rate an overall best response of either complete response (CR) or partial response (PR) by local assessment. CR was defined as the disappearance of all target lesions and reduction in short axis of any pathologic lymphnode to <10 mm. PR was defined as ≥3 0% decrease in the sum of diameters of target lesions, taking the baseline sum diameters. Per planned analysis, ORR by Local Assessment was assessed for TNBC Target Population, HR+/HER2-mBC Population, and mUC Population.
Time Frame: Up to data cutoff date of 01 March 2019 (maximum duration: 74 months)
Population: * Target mTNBC: Participants with mTNBC who received at least 2 prior therapies for metastatic disease & who received at least 1 dose of 10 mg/kg SG
  * HR+/HER2-mBC: Participants with HR+/HER2- mBC who progressed on at least 1 prior hormonal therapy & who received at least 1 dose of 10 mg/kg SG
  * mUC: Participants who had relapsed after or were refractory to at least 1 prior treatments & who received at least 1 dose of 10 mg/kg SG
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TNBC Target Population | HR+/HER2- mBC Population | mUC Population
Number analyzed (Participants) | 108 | 54 | 45
Percentage of participants | 33.3 [24.6 to 43.1] | 31.5 [19.5 to 45.6] | 28.9 [16.4 to 44.3]

6. Secondary Outcome: Duration of Response by ICR
Description: Duration of Response was defined as the duration of overall response measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Per planned analysis, ORR by ICR was assessed for the TNBC Target Population only.
Time Frame: Up to data cutoff date of 01 March 2019 (maximum duration: 74 months)
Population: Target mTNBC: Participants with mTNBC who received at least 2 prior therapies for metastatic disease and who received SG at a dose of 10 mg/kg. Per planned analysis, ORR by ICR was assessed for the TNBC Target Population only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TNBC Target Population
Number analyzed (Participants) | 108
months | 9.1 [4.6 to 11.3]

7. Secondary Outcome: Duration of Response by Local Assessment
Description: Duration of Response was defined as the duration of overall response measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Per planned analysis, duration of response by local assessment was assessed for TNBC Target Population, HR+/HER2-mBC Population, and mUC Population.
Time Frame: Up to data cutoff date of 01 March 2019 (maximum duration: 74 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TNBC Target Population | HR+/HER2- mBC Population | mUC Population
Number analyzed (Participants) | 108 | 54 | 45
months | 7.7 [4.9 to 10.8] | 8.7 [3.7 to 12.7] | 12.9 [3.8 to 22.5]

8. Secondary Outcome: Time to Response by ICR
Description: Time to response was defined as the time from the first dose to the first documentation of response (PR or CR). Per planned analysis, time to response by ICR was assessed for the TNBC Target Population only.
Time Frame: Up to data cutoff date of 01 March 2019 (maximum duration: 74 months)
Population: Target mTNBC: Participants with mTNBC who received at least 2 prior therapies for metastatic disease & who received at least 1 dose of 10 mg/kg SG
Measure: Median (Full Range); unit: months
Arm/Group | TNBC Target Population
Number analyzed (Participants) | 108
months | 2.2 [1.6 to 7.6]

9. Secondary Outcome: Time to Response by Local Assessments
Description: Time to response was defined as the time from the first dose to the first documentation of response (PR or CR). Per planned analysis, time to response by local assessment was assessed for TNBC Target Population, HR+/HER2-mBC Population, and mUC Population.
Time Frame: Up to data cutoff date of 01 March 2019 (maximum duration: 74 months)
Population: as for outcome 5
Measure: Median (Full Range); unit: months
Groups:
- TNBC Target Population (TNBC Population): Overall 144 participants with TNBC were enrolled in the study and received at least one dose of SG. Of these 144 participants, 108 received at least 2 prior therapies for metastatic disease and were treated with SG at a starting dose of 10mg/kg. These 108 participants were included in the analysis of safety and were referred to as the TNBC Target Population.
- HR+/HER2- mBC Population (Non-TNBC): Overall 68 participants with non-TNBC were enrolled in the study and received at least one dose of SG. Of these 68 participants, 54 were confirmed as HR+/HER2-, had progressed on at least one prior hormonal therapy in the metastatic setting, and had received at least one dose of 10 mg/kg SG. These 54 participants were included in the analysis of safety and were referred to as the HR+/HER2- mBC Population.
Arm/Group | TNBC Target Population (TNBC Population) | HR+/HER2- mBC Population (Non-TNBC) | mUC Population
Number analyzed (Participants) | 108 | 54 | 45
months | 2.0 [1.6 to 13.5] | 2.1 [1.4 to 7.8] | 1.9 [1.7 to 7.4]

10. Secondary Outcome: Clinical Benefit Rate (CBR) by Local Assessment
Description: Clinical benefit rate (CR+PR+[stable disease (SD) ≥ 6 months]) is defined as those participants with best response as CR or PR or else SD with a duration of at least 6 months. SD for 6 months duration was defined as the time from the first dose to the first documentation of PD or to the last adequate response assessment prior to data cut-off date, whichever is earlier. Per planned analysis, CBR by local assessment was assessed for TNBC Target Population, HR+/HER2-mBC Population, and mUC Population.
Time Frame: Up to data cutoff date of 01 March 2019 (maximum duration: 74 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TNBC Target Population | HR+/HER2- mBC Population | mUC Population
Number analyzed (Participants) | 108 | 54 | 45
Percentage of participants | 45.4 [35.8 to 55.2] | 44.4 [30.9 to 58.6] | 44.4 [29.6 to 60.0]

11. Secondary Outcome: Progression Free Survival (PFS) by Local Assessment
Description: Progression-free survival (PFS) was defined as the interval from the first dose start date to the date of disease progression defined as documented progressive disease (PD) or death from any cause, whichever occurs first. Per planned analysis, PFS by local assessment was assessed for TNBC Target Population, HR+/HER2-mBC Population, and mUC Population.
Time Frame: Up to data cutoff date of 01 March 2019 (maximum duration: 74 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TNBC Target Population | HR+/HER2- mBC Population | mUC Population
Number analyzed (Participants) | 108 | 54 | 45
months | 5.6 [4.8 to 6.6] | 5.5 [3.6 to 7.6] | 6.8 [3.6 to 9.7]

12. Secondary Outcome: Overall Survival by Local Assessment
Description: Overall survival was defined as the time from the date of the first dose start date to the date of death due to any cause. Per planned analysis, overall survival by local assessment was assessed for TNBC Target Population, HR+/HER2-mBC Population, and mUC Population.
Time Frame: Up to data cutoff date of 01 March 2019 (maximum duration: 74 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Groups:
- HR+/HER2- mBC Population: Overall, 68 participants with non-TNBC were enrolled in the study and received at least one dose of SG. Of these 68 participants, 54 were confirmed as HR+/HER2-, had progressed on at least one prior hormonal therapy in the metastatic setting, and had received at least one dose of 10 mg/kg SG. These 54 participants were included in the analysis of safety and were referred to as the HR+/HER2- mBC Population.
Arm/Group | TNBC Target Population | HR+/HER2- mBC Population | mUC Population
Number analyzed (Participants) | 108 | 54 | 45
months | 13.0 [11.2 to 14.0] | 12.0 [9.0 to 18.2] | 16.8 [9.0 to 21.9]

13. Secondary Outcome: Pharmacokinetic (PK) Parameter: T1/2 of Total Antibody, SN-38 Glucuronide, Total SN-38, Sacituzumab Govitecan-hziy, and Free SN-38
Description: T1/2 was determined for 5 analytes: total antibody, SN-38 glucuronide, total SN-38, free SN-38, and sacituzumab govitecan-hziy, a derived antibody drug conjugate (ADC) concentration. SN-38 is one of the components of sacituzumab govitecan-hziy. T1/2 is defined as apparent terminal elimination half-life (h); calculated as 0.693/λz. The dose level evaluated for PK analysis was 10 mg/kg.
Time Frame: Cycle 1: Preinfusion, 30 minutes and 3-4 hours post infusion, then 1 day, 2 days, 3 days, and 7 days later (1 Cycle = 21 days). Infusion duration: 3 hours (± 30 minutes) for 1st infusion; 1-2 hours (± 30 minutes) for subsequent infusions
Population: Participants with epithelial cancer that involved any one of the following with available data were analyzed: cervical cancer, colorectal cancer, endometrial cancer, epithelial ovarian cancer, esophageal cancer, gastric adenocarcinoma, glioblastoma multiforme, head & neck cancers- squamous cell, hepatocellular carcinoma, hormone-refractory prostate cancer, metastatic, non-small-cell lung cancer, pancreatic ductal adenocarcinoma, renal cell cancer, small-cell lung cancer, non TNBC, TNBC and mUC.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Groups:
- SG 10 mg/kg: Participants included adults with the following tumor types:
  cervical cancer, colorectal cancer, endometrial cancer, epithelial ovarian cancer, esophageal cancer, gastric adenocarcinoma, glioblastoma multiforme, head and neck cancers- squamous cell, hepatocellular carcinoma, hormone-refractory prostate cancer, metastatic, non-small-cell lung cancer, pancreatic ductal adenocarcinoma, renal cell cancer, small-cell lung cancer, non-triple-negative breast cancer, triple-negative breast cancer, and metastatic urothelial cancer.
  All participants received SG 10 mg/kg of body weight by IV infusion on Days 1 and 8 of a 21-day treatment cycle.
Arm/Group | SG 10 mg/kg
Number analyzed (Participants) | 128
hours
  Total Antibody: number analyzed (Participants) | 5
  Total Antibody | 66.6 (14.4)
  SN-38G: number analyzed (Participants) | 63
  SN-38G | 21.4 (24.5)
  Total SN-38 | 20.2 (26.6)
  Sacituzumab Govitecan-hziy (SG): number analyzed (Participants) | 120
  Sacituzumab Govitecan-hziy (SG) | 15.0 (15.3)
  Free SN-38: number analyzed (Participants) | 95
  Free SN-38 | 17.1 (18.6)

14. Secondary Outcome: PK Parameter: AUC0-24 of Total Antibody, SN-38 Glucuronide, Total SN-38, Sacituzumab Govitecan-hziy, and Free SN-38
Description: AUC0-24 was determined for 5 analytes: total antibody, SN-38 glucuronide, total SN-38, free SN-38, and sacituzumab govitecan-hziy, a derived antibody drug conjugate (ADC) concentration. SN-38 is one of the components of sacituzumab govitecan-hziy. AUC0-24 is defined as area under the serum concentration-time curve from time 0 to 24 hours. The dose level evaluated for PK analysis was 10 mg/kg.
Time Frame: Cycle 1: Preinfusion, 30 minutes and 3-4 hours post infusion, then 1 day, 2 days, 3 days, and 7 days later (1 Cycle = 21 days). Infusion duration: 3 hours (± 30 minutes) for 1st infusion; 1-2 hour (± 30 minutes) for subsequent infusions
Population: Participants with epithelial cancer that involved any one of the following with available data were analyzed: cervical cancer, colorectal cancer, endometrial cancer, epithelial ovarian cancer, esophageal cancer, gastric adenocarcinoma, glioblastoma multiforme, head & neck cancers- squamouse cell, hepatocellular carcinoma, hormone-refractory prostate cancer, metastatic, non-small-cell lung cancer, pancreatic ductal adenocarcinoma, renal cell cancer, small-cell lung cancer, non TNBC, TNBC and mUC.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per liter
Arm/Group | SG 10 mg/kg
Number analyzed (Participants) | 128
microgram*hour per liter
  Total Antibody: number analyzed (Participants) | 5
  Total Antibody | 4940 (30.1)
  SN-38G: number analyzed (Participants) | 63
  SN-38G | 0.370 (45.6)
  Total SN-38 | 65.5 (29.2)
  Sacituzumab Govitecan-hziy (SG): number analyzed (Participants) | 120
  Sacituzumab Govitecan-hziy (SG) | 3290 (25.2)
  Free SN-38: number analyzed (Participants) | 95
  Free SN-38 | 1.67 (58.5)

15. Secondary Outcome: PK Parameter: AUC0-168 of Total Antibody, SN-38 Glucuronide, Total SN-38, Sacituzumab Govitecan-hziy, and Free SN-38
Description: AUC0-168 was determined for 5 analytes: total antibody, SN-38 glucuronide, total SN-38, free SN-38, and sacituzumab govitecan-hziy, a derived antibody drug conjugate (ADC) concentration. SN-38 is one of the components of sacituzumab govitecan-hziy. AUC0-168 is defined as area under the serum concentration-time curve from time 0 to 168 hours. The dose level evaluated for PK analysis was 10 mg/kg.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per liter
Arm/Group | SG 10 mg/kg
Number analyzed (Participants) | 128
microgram*hour per liter
  Total Antibody: number analyzed (Participants) | 5
  Total Antibody | 20800 (22.2)
  SN-38G: number analyzed (Participants) | 63
  SN-38G | 0.842 (50.0)
  Total SN-38 | 107 (25.4)
  Sacituzumab Govitecan-hziy (SG): number analyzed (Participants) | 120
  Sacituzumab Govitecan-hziy (SG) | 5050 (24.4)
  Free SN-38: number analyzed (Participants) | 95
  Free SN-38 | 3.08 (56.6)

16. Secondary Outcome: PK Parameter: AUC0-inf of Total Antibody, SN-38 Glucuronide, Total SN-38, Sacituzumab Govitecan-hziy, and Free SN-38
Description: AUC0-inf was determined for 5 analytes: total antibody, SN-38 glucuronide, total SN-38, free SN-38, and sacituzumab govitecan-hziy, a derived antibody drug conjugate (ADC) concentration. SN-38 is one of the components of sacituzumab govitecan-hziy. AUC0-inf is defined as area under the serum concentration-time curve from time 0 extrapolated to infinity. The dose level evaluated for PK analysis was 10 mg/kg.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per liter
Arm/Group | SG 10 mg/kg
Number analyzed (Participants) | 128
microgram*hour per liter
  Total Antibody: number analyzed (Participants) | 5
  Total Antibody | 25100 (20.5)
  SN-38G: number analyzed (Participants) | 63
  SN-38G | 0.850 (50.7)
  Total SN-38 | 107 (25.5)
  Sacituzumab Govitecan-hziy (SG): number analyzed (Participants) | 120
  Sacituzumab Govitecan-hziy (SG) | 5050 (24.4)
  Free SN-38: number analyzed (Participants) | 95
  Free SN-38 | 3.08 (56.6)

17. Secondary Outcome: PK Parameter: Cmax of Total Antibody, SN-38 Glucuronide, Total SN-38, Sacituzumab Govitecan-hziy, and Free SN-38
Description: Cmax was determined for 5 analytes: total antibody, SN-38 glucuronide, total SN-38, free SN-38, and sacituzumab govitecan-hziy, a derived antibody drug conjugate (ADC) concentration. SN-38 is one of the components of sacituzumab govitecan-hziy. Cmax is defined as maximum observed serum concentration obtained directly from the observed concentration-time data. The dose level evaluated for PK analysis was 10 mg/kg.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter
Arm/Group | SG 10 mg/kg
Number analyzed (Participants) | 128
microgram per liter
  Total Antibody: number analyzed (Participants) | 5
  Total Antibody | 245 (26.9)
  SN-38G: number analyzed (Participants) | 63
  SN-38G | 0.0206 (50.4)
  Total SN-38 | 4.39 (25.2)
  Sacituzumab Govitecan-hziy (SG): number analyzed (Participants) | 120
  Sacituzumab Govitecan-hziy (SG) | 220 (24.7)
  Free SN-38: number analyzed (Participants) | 95
  Free SN-38 | 0.0992 (61.1)

ADVERSE EVENTS:
Time Frame: - Adverse Events: First dose date up to 91.88 months plus 30 days - All-Cause Mortality: First dose date up to 91.88 months
Description: Overall Safety Population: All participants who received at least 1 dose of SG. Per planned analysis, data were collected for the Overall Safety Population, pooling all participants regardless of dose level received.
Groups:
- Overall Safety Population: All participants who were enrolled in the study and received one dose of sacituzumab govitecan-hziy (SG) at dose level of either 8 mg/kg, 10 mg/kg, 12 mg/kg, or 18 mg/kg of body weight via intravenous (IV) infusion on Days 1 and 8 of a 21-day treatment cycle until disease progression or unacceptable toxicity.
Arm/Group | Overall Safety Population
All-Cause Mortality (participants affected / at risk) | 422/495
Serious Adverse Events (participants affected / at risk) | 192/495
Other Adverse Events (participants affected / at risk) | 490/495
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Safety Population (N=495)
Anaemia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 20
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 7
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Cardiac tamponade (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Purtscher retinopathy (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 18
Dysphagia (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 10
Neutropenic colitis (Gastrointestinal disorders) | 2
Oesophageal obstruction (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pouchitis (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 7
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 11
Asthenia (General disorders) | 3
Chest pain (General disorders) | 4
Face oedema (General disorders) | 1
Fatigue (General disorders) | 4
Gait disturbance (General disorders) | 1
Generalised oedema (General disorders) | 2
Localised oedema (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 5
Pyrexia (General disorders) | 4
Systemic inflammatory response syndrome (General disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Anaphylactic reaction (Immune system disorders) | 1
Clostridium difficile colitis (Infections and infestations) | 2
Clostridium difficile infection (Infections and infestations) | 1
Covid-19 pneumonia (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Epiglottitis (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pleural infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 14
Pyelonephritis (Infections and infestations) | 1
Rectal abscess (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Septic shock (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Vascular device infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Post procedural fever (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 4
Failure to thrive (Metabolism and nutrition disorders) | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Vocal cord paralysis (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 2
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 4
Acute kidney injury (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Urinary tract obstruction (Renal and urinary disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Vocal cord dysfunction (Respiratory, thoracic and mediastinal disorders) | 1
Paraneoplastic dermatomyositis (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Embolism (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Peripheral embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Safety Population (N=495)
Anaemia (Blood and lymphatic system disorders) | 207
Neutropenia (Blood and lymphatic system disorders) | 196
Abdominal distension (Gastrointestinal disorders) | 25
Abdominal pain (Gastrointestinal disorders) | 108
Constipation (Gastrointestinal disorders) | 184
Diarrhoea (Gastrointestinal disorders) | 303
Dyspepsia (Gastrointestinal disorders) | 26
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 25
Nausea (Gastrointestinal disorders) | 342
Stomatitis (Gastrointestinal disorders) | 27
Vomiting (Gastrointestinal disorders) | 220
Asthenia (General disorders) | 27
Chest pain (General disorders) | 33
Chills (General disorders) | 33
Fatigue (General disorders) | 280
Oedema peripheral (General disorders) | 79
Pain (General disorders) | 27
Pyrexia (General disorders) | 80
Upper respiratory tract infection (Infections and infestations) | 60
Urinary tract infection (Infections and infestations) | 65
Activated partial thromboplastin time prolonged (Investigations) | 33
Alanine aminotransferase increased (Investigations) | 44
Aspartate aminotransferase increased (Investigations) | 47
Blood alkaline phosphatase increased (Investigations) | 55
Lymphocyte count decreased (Investigations) | 38
Neutrophil count decreased (Investigations) | 98
Weight decreased (Investigations) | 75
White blood cell count decreased (Investigations) | 77
Decreased appetite (Metabolism and nutrition disorders) | 171
Dehydration (Metabolism and nutrition disorders) | 78
Hyperglycaemia (Metabolism and nutrition disorders) | 54
Hypoalbuminaemia (Metabolism and nutrition disorders) | 30
Hypocalcaemia (Metabolism and nutrition disorders) | 26
Hypokalaemia (Metabolism and nutrition disorders) | 89
Hypomagnesaemia (Metabolism and nutrition disorders) | 89
Hyponatraemia (Metabolism and nutrition disorders) | 38
Hypophosphataemia (Metabolism and nutrition disorders) | 65
Arthralgia (Musculoskeletal and connective tissue disorders) | 68
Back pain (Musculoskeletal and connective tissue disorders) | 75
Muscular weakness (Musculoskeletal and connective tissue disorders) | 31
Myalgia (Musculoskeletal and connective tissue disorders) | 28
Pain in extremity (Musculoskeletal and connective tissue disorders) | 45
Dizziness (Nervous system disorders) | 81
Dysgeusia (Nervous system disorders) | 33
Headache (Nervous system disorders) | 78
Neuropathy peripheral (Nervous system disorders) | 30
Anxiety (Psychiatric disorders) | 30
Depression (Psychiatric disorders) | 29
Insomnia (Psychiatric disorders) | 57
Haematuria (Renal and urinary disorders) | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 101
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 100
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 32
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 29
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 40
Alopecia (Skin and subcutaneous tissue disorders) | 216
Dry skin (Skin and subcutaneous tissue disorders) | 38
Pruritus (Skin and subcutaneous tissue disorders) | 62
Rash (Skin and subcutaneous tissue disorders) | 78
Hypotension (Vascular disorders) | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Immunomedics, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Immunomedics in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT01631552/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT01631552/SAP_001.pdf